CLINICAL TRIAL: NCT06851299
Title: Randomized Controlled Clinical Study of Efficacy and Safety of Trop2-ADC Monotherapy or Combination Immunotherapy Strategies in the Treatment of Advanced Triple-negative Breast Cancer
Brief Title: The Clinical Study of the Efficacy and Safety of Trop2-ADC Monotherapy or Combination Immunotherapy Strategy in the Treatment of Advanced Triple-negative Breast Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2025-007-02
Record Dates: First submitted 2025-02-11; First posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — arginine decarboxylase

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Accept ADC monotherapy (Active Comparator)
  Interventions: Drug: trop2-ADC
- Accept ADC combined with anti-angiogenic drug (Experimental)
  Interventions: Drug: ADC +anti-angiogenic drug
- Receive ADC in combination with PD1 monoclonal antibody and anti-angiogenic drug (Experimental)
  Interventions: Drug: ADC + PD1 monoclonal antibody +anti-angiogenic drug

INTERVENTIONS:
Drug: trop2-ADC — Accept ADC monotherapy
  Arms: Accept ADC monotherapy
Drug: ADC +anti-angiogenic drug — Accept ADC combined with anti-angiogenic drug
  Arms: Accept ADC combined with anti-angiogenic drug
Drug: ADC + PD1 monoclonal antibody +anti-angiogenic drug — ADC combined with PD1 monoclonal antibody and anti-angiogenic drug
  Arms: Receive ADC in combination with PD1 monoclonal antibody and anti-angiogenic drug

SUMMARY:
This is a prospective, multicenter, randomized controlled study aimed at evaluating the efficacy and safety of Trop2-ADC monotherapy or immune combination strategy in the treatment of advanced triple-negative breast cancer.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized controlled study aims to evaluate the 3-month treatment efficacy (ORR) of three therapeutic strategies-ADC monotherapy, ADC in combination with immunotherapy, and ADC in combination with immunotherapy and anti-angiogenesis-in patients with advanced breast cancer, and to assess potential adverse events related to the treatment regimens. Participants will receive treatment with a Trop-2-targeting ADC drug containing a TOP1 inhibitor (such as Gosituzumab or SKB264), in accordance with the defined protocol. Regular assessments will include imaging, histopathological analysis, and safety monitoring. The objective of this study is to provide novel treatment strategies for triple-negative breast cancer by evaluating the efficacy and safety of trop2-ADC+ immunotherapy + antiangiogenic agents and trop2-ADC+ antiangiogenic agents versus trop2-ADC monotherapy in patients with metastatic triple-negative breast cancer (mTNBC).

ELIGIBILITY:
Inclusion Criteria:

* 1) adult female patients (aged 18-70 years) with metastatic triple negative breast cancer confirmed by pathology or imaging;
* 2) no more than two previous lines of therapy for metastatic disease;
* 3) ECOG performance status ≤2 and expected survival time ≥ 3 months;
* 4) At least one measurable lesion on imaging within 2 weeks before enrollment; Or simple bone metastases;
* 5) Prior treatment-related toxicity at enrollment had to be resolved to NCI CTCAE version 5.0 ≤ grade 1 (excluding alopecia or any other toxicity deemed by the investigator to be of no risk to patient safety)
* 6) adequate bone marrow reserve: a. White blood cell count (WBC) ≥3.0×10^9 / L, b. Neutrophil count (ANC) ≥1.5×10^9 / L, c. Platelet count (PLT) ≥70×10^9 / L
* 7) liver, kidney and heart function tests were basically normal (according to the normal values of the laboratories in the study center) : a. Total bilirubin (TBIL) ≤3× upper limit of normal value (ULN), b. alanine aminotransferase and aspartate aminotransferase (ALT/AST) ≤2.5×ULN (≤5xULN in patients with liver metastases), c. Total bilirubin (TBIL) ≤3× upper limit of normal value (ULN), B. alanine aminotransferase and aspartate aminotransferase (Alt /AST) ≤2.5×ULN (≤5xULN in patients with liver metastases). Serum creatinine ≤1.5×ULN or creatinine clearance (Ccr) ≥60 ml/min; d. Left ventricular ejection fraction (LVEF) ≥ 55%, e. QTcF(Fridericia correction) ≤ 470 ms.
* 8) understood the study process and volunteered to participate in the study. Informed consent was signed.

Exclusion Criteria:

* 1) patients with a known allergy to the active ingredient or other ingredient of the study drug.
* 2) patients with known resistance to trop2-ADC drugs. 、
* 3) receiving radiotherapy, chemotherapy, or endocrine therapy within 4 weeks before enrollment, or participating in any interventional drug clinical trial;
* 4) pregnant or lactating women or women of childbearing age who refused to use effective contraception during the study period.
* 5) patients with severe cardiac disease or discomfort expected to be unable to tolerate chemotherapy, including but not limited to: fatal arrhythmia or higher grade atrioventricular block, unstable angina pectoris, clinically significant valvular heart disease, transmural myocardial infarction on ECG, uncontrolled hypertension;
* 6) any other condition considered by the investigator to be inappropriate for participation in the study, a concomitant disease or condition that could interfere with participation in the study, or any serious medical disorder that could affect the safety of the subject (e.g., uncontrolled heart disease, hypertension, active or uncontrolled infection, active hepatitis B virus infection)；

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Objective response rate 3 months after treatment (ORR) | Three months after enrollment

SECONDARY OUTCOMES:
Overall survival (OS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
living quality | "through study completion, an average of 1 year
  The scores of EORTC-c30 scale were compared before and after enrollment.
Clinical benefit rate | 3 months after enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Tumor Center, Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, China;, Guangzhou, Guangdong, China